CLINICAL TRIAL: NCT01467544
Title: Exploring the Effects of Tai Chi on Cardiometabolic Risk in Women
Brief Title: Reduce Cardiovascular Risk in Women Through Tai Chi Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13605; P30NR011403 (NIH)
Record Dates: First submitted 2011-10-27; First posted 2011-11-08 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Cardiometabolic Risk; Cardiovascular Disease
Keywords: Tai Chi
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wait list control group (No Intervention): After completing time three data collection, wait-listed participants will be provided with the complete tai chi intervention (8 weeks).
- Tai Chi intervention group (Experimental): This participant group completes the 8-week tai chi group intervention.
  Interventions: Other: Tai Chi class

INTERVENTIONS:
Other: Tai Chi class — The 8-week tai chi group intervention will be lead by Project PI. A focused short form of tai chi involving 12 movements will be used in this project. Each of 8 weekly 60-minute sessions will begin with a 10-minute guided meditation session. Movements learned the previous week will be reviewed prior to introducing new movements. Training DVDs will be produced and provided to participants for weekly and ongoing practice of the techniques.
  Arms: Tai Chi intervention group

SUMMARY:
Tai chi intervention may lead to relaxation and could potentially reduce the risk of cardiovascular disease. This project entails a comprehensive and innovative approach for understanding, measuring, and potentially reducing cardiovascular risk in women. The goal of this area of research is to reduce cardiovascular risk and perhaps reduce illness and death.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the United States. Historically, CVD has been under diagnosed and inadequately treated in women related to issues of gender bias, lack of public and medical awareness of its prevalence, and its unique presenting symptomatology. Despite increasing awareness, as well as better diagnostics and treatment, women are still more likely than men to present with advanced disease and experience higher CVD-related morbidity and mortality. Given these facts, prevention of CVD is critical. Cardiometabolic risk (CMR) is a relatively new term for a set of risk factors that, when viewed together, are indicators of overall risk for developing CVD. CMR is useful for assessing, modifying, and ultimately preventing the development of CVD. Prevention of CVD in women may best be achieved by early identification and treatment of evolving CMR. Central or abdominal obesity, reflecting the presence of visceral adipose tissue and evidenced by increased waist circumference, has been shown to be a significant predictor of CVD. In this PNI-based model of CMR and fatigue, abdominal adiposity and fatigue are products of allostatic load. Resulting from cumulative wear and tear, fatigue gives rise to dysregulation of metabolic processes, ultimately resulting in subjective symptomatology and disease risk. Additionally, fatigue often accompanies metabolic changes, potentiating a trajectory of CMR related to decreased physical activity and self-care. Tai chi may enhance relaxation and could potentially reduce CMR. The specific aims of this project are to refine a tai chi intervention using a wait-list pretest-posttest design with repeated measures. Feasibility and acceptability of the intervention and identification of potential indicators of effectiveness also will be assessed. Additionally, a PNI-based model of fatigue and CMR will be further refined. The first aim will be analyzed using a mixed effects model. The second specific aim, to refine a PNI-based model of fatigue and CMR, will be examined using descriptive statistics, graphical methods and pairwise correlations and, as a second step, variable reduction methods including factor analysis, principle component analysis and canonical correlation analysis. The project is based on a theoretically and scientifically sound framework to investigate a more comprehensive, sensitive, and innovative model for understanding, measuring, and potentially reducing CMR in women. With further studies, the goal of this line of research is to reduce CMR and perhaps reduce morbidity and mortality related to CVD.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women
* able to read and speak English
* self-reported histories of CVD in first- or second-degree relatives

Exclusion Criteria:

* previous diagnosis of CVD, DM, uncontrolled or severe hypertension (defined as >180/120),
* LDL-C greater than or equal to 160,
* fasting blood glucose greater than or equal to 126,
* morbid obesity (BMI > 40), or
* unstable major depressive disorder.
* taken corticosteroids within 30 days and 72 hours of inhaled or nasal steroids of data collection.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the intervention | 8weeks intervention & post-class focus group

SECONDARY OUTCOMES:
Identify potential indicators of intervention effectiveness (change in PNI measures). | baseline
Identify potential indicators of intervention effectiveness (change in PNI measures). | 8 Weeks
Identify potential indicators of intervention effectiveness (change in PNI measures). | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lynne W Robins, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States